CLINICAL TRIAL: NCT00210847
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Tramadol HCl/Acetaminophen for the Treatment of Painful Diabetic Neuropathy
Brief Title: A Study Comparing the Effectiveness and Safety of Tramadol HCl/Acetaminophen Versus Placebo for the Treatment of Painful Neuropathy in Diabetic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004660
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Diabetic Neuropathies
Keywords: peripheral neuropathy; Diabetic neuropathy; pain; diabetes; extremities; neuropathy; diabetic
MeSH Terms: conditions — Diabetic Neuropathies; Peripheral Nervous System Diseases; Pain; Diabetes Mellitus | interventions — Ultracet

INTERVENTIONS:
Drug: tramadol, acetaminophen

SUMMARY:
The purpose of this study is to explore the pain-reieiving effects and safety of tramadol HCl/acetaminophen as compared to placebo in patients experiencing painful diabetic neuropathy. Treatment of neuropathic pain often requires the use of more than one medication. The pain-relieving potential of tramadol HCl/acetaminophen for the treatment of painful diabetic neuropathy comes from the multiple mechanisms of action in this combination pain medication. Patients who experience painful diabetic neuropathy will be enrolled in this study.

DETAILED DESCRIPTION:
Previous studies have shown that tramadol HCl is effective in painful diabetic neuropathy. The treatment of neuropathic pain often requires the use of more than one medication, working through different mechanisms of action, to provide the best pain relief. The pain-relieving potential of tramadol HCl /acetaminophen for the treatment of painful diabetic neuropathy comes from the multiple mechanisms of action in this combination pain medication. This is a multicenter, randomized, double-blind, placebo-controlled, parallel group study. Patients who experience painful diabetic neuropathy will be enrolled. There will be a period of up to 3 weeks during which patients will stop taking medications not allowed by the study. A 7-day baseline period will follow, during which time patients will call into an Interactive Voice Response (IVR) system every night at bedtime to record daily assessments including average daily pain and sleep interference. Patients who enter the double-blind portion of the study will be randomized (like with the toss of a coin) to receive either tramadol HCl/acetaminophen or placebo. The dose of tramadol HCl/acetaminophen or placebo will be gradually increased until the doctor determines the patient is taking an adequate dose; up to 1 or 2 tablets 4 times per day, but not more than 8 tablets per day. Every night at bedtime during the double-blind phase, patients will call the IVR system to report assessments of average daily pain, sleep interference and the number of tablets of study medication taken that day. At the end of the study, patients will be tapered off their study medication. The objective of this study is to compare the analgesic effectiveness and safety of tramadol HCl/acetaminophen versus placebo for the treatment of painful diabetic neuropathy.

1 or 2 tramadol HCl (37.5 milligrams)/acetaminophen (325 milligrams) combination tablets or matching placebo by mouth up to 4 times a day for 66 days

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetic neuropathy in both lower extremities
* Lower extremity pain for at least 3 months
* Stable treatment of diabetes with drugs or diet for at least 3 months
* Documented history of Type I or II diabetes with current treatment control (glycosylated hemoglobin A1c of <10%)
* Documented daily pain on at least 4 of 7 days during baseline period (pain rated at least 5 on scale of 11)
* In generally good health
* If female of childbearing potential, using acceptable method of birth control

Exclusion Criteria:

* No failed trials of tramadol HCl or tramadol HCl/acetaminophen
* No participation in more than 2 clinical trials for treatment of neuropathic pain
* No more than 2 failed trials of medications for neuropathic pain
* No use of prohibited concomitant medications
* No peripheral neuropathy caused by condition other than diabetes
* No other pain more severe than neuropathic pain
* No progressive or degenerative neurological disorder
* No painful peripheral diabetic neuropathy for > 10 years
* No kidney or liver dysfunction
* Not pregnant or breast-feeding
* No unstable medical disease
* No clinically significant medical conditions
* No condition that might affect the way the body absorbs or processes the study drug
* No history of suicide attempt/tendencies
* No major psychiatric disorder in past 6 months
* No history of drug or alcohol abuse/dependance in the past 2 years
* No amputations
* No active infection of the lower extremity
* No active foot ulcer
* No use of an investigational drug in past 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2003-12; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Change in the average of daily pain score recorded in the IVR system from baseline to the patient's final week of treatment with study medication.

SECONDARY OUTCOMES:
Efficacy measured by Brief Pain Inventory, Visual Analogue Scale, Short-Form McGill Pain Questionnaire, Profile of Mood States, SF-36 Health Survey, Physician and Subject Global Impression of Change, average daily sleep interference

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Freeman R, Raskin P, Hewitt DJ, Vorsanger GJ, Jordan DM, Xiang J, Rosenthal NR; CAPSS-237 Study Group. Randomized study of tramadol/acetaminophen versus placebo in painful diabetic peripheral neuropathy. Curr Med Res Opin. 2007 Jan;23(1):147-61. doi: 10.1185/030079906X162674. PMID 17257476
- See also: Clinical Study Report: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Tramadol HCl/Acetaminophen for the Treatment of Painful Diabetic Neuropathy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=615&filename=CR004660_CSR.pdf